CLINICAL TRIAL: NCT00481728
Title: Evaluation of Sympathetic Skin Responses and Heart Rate Variability as Objective Measures of Bladder Sensation - a Double Blind Third Party Open Placebo Controlled Randomised Study Using a Single Dose of Tolterodine in Patients With Idiopathic Overactive Bladder and Healthy Volunteers
Brief Title: Evaluation of the Link Between Bladder Sensation and Changes in Skin Electrical Conductance and Heart Rate.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: A6121189
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Tolterodine (Experimental)
  Interventions: Drug: Tolterodine; Procedure: Filling cystometry; Procedure: Intravesical neurostimulation

INTERVENTIONS:
Drug: Tolterodine — Single dose per patient as determined by protocol.
Procedure: Filling cystometry — This is a procedure.
Procedure: Intravesical neurostimulation — This is a procedure.

SUMMARY:
Measuring sympathetic skin response or heart rate variability can provide an objective biomarker of bladder sensation and its modulation by drug with potential to treat overactive bladder.

DETAILED DESCRIPTION:
Evaluation of the link between bladder sensation and changes in skin electrical conductance and heart rate.

ELIGIBILITY:
Inclusion Criteria:

* Female, healthy volunteers or OAB patients 18-65 years old, non pregnant and non lactating

Exclusion Criteria:

* History of lower urinary tract pathology
* Excessive alcohol and tobacco consumption
* Treatment with investigational drug in the last 30 days
* Abnormal ECG trace
* Conditions that would contraindicate the use of tolterodine or any other anti muscarinic agent

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Heart rate variability evoked by filling cystometry and intravesical neurostimulation and sympathetic skin response evoked by intravesical neurostimulation in healthy volunteers and OAB patients

SECONDARY OUTCOMES:
To investigate the correlation between the changes in heart rate variability and sympathetic skin response evoked by filling cystometry and intravesical neurostimulation in OAB patients. | duration of study
To determine whether there is a difference in the stimulus response relationship for the evoked changes in HRV and SSR between healthy volunteers and OAB patients. | duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Zurich, Switzerland

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6121189&StudyName=Evaluation%20of%20the%20link%20between%20bladder%20sensation%20and%20changes%20in%20skin%20electrical%20conductance%20and%20heart%20rate.